CLINICAL TRIAL: NCT01240083
Title: Effectiveness of Theta-burst Stimulation (TBS) Versus Tonic High Frequency Repetitive Transcranial Magnetic Stimulation (rTMS)in Patients With Major Depression
Brief Title: Effectiveness of Theta-burst Stimulation (TBS) in Patients With Major Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Berthold Langguth, MD, Ph.D., MD, Ph.D., University of Regensburg
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Uni-Reg-TB1
Record Dates: First submitted 2010-11-12; First posted 2010-11-15 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Depression
Keywords: Depression; Transcranial magnetic stimulation; Thetaburst Stimulation; Alternative treatment methods
MeSH Terms: conditions — Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Thetaburst Stimulation (Experimental): 1: Thetaburst stimulation: right DLPFC continuous TBS followed by left DLPFC intermitted TBS each with 50 Hz, together 1200 stimuli, 80% motorthreshold
  Interventions: Device: Thetaburst Stimulation
- High frequency rTMS (Experimental): 2: Experimental high frequency rTMS ( Alpine Biomed Mag Pro Option) : 1000 stimuli of 1 Hz over the right DLPFC, 110% motor threshold, followed by 1000 stimuli of 10 Hz over the left DLPFC , 110% motorthreshold
  Interventions: Device: High frequency rTMS
- Placebo Stimulation (Experimental): 3: Sham Stimulation (Sham coil): right DLPFC continuous TBS, followed by left DLPFC intermitted TBS each with 50 Hz, together 1200 Stimuli, 80% motorthreshold
  Interventions: Device: Placebo Stimulation

INTERVENTIONS:
Device: Thetaburst Stimulation — Thetaburst stimulation: continuous TBS over the right DLPFC, followed by intermitted TBS over the left DLPFC, each with 50 Hz, together 1200 stimuli (80% motorthreshold)
  Other Names: Transcranial Magnetic Stimulation; Theta-burst
  Arms: Thetaburst Stimulation
Device: High frequency rTMS — Experimental high frequency rTMS ( Alpine Biomed Mag Pro Option) : 1000 stimuli of 1 Hz over the right DLPFC (110% motor threshold)followed by 1000 stimuli of 10 Hz over the left DLPFC (110% motorthreshold)
  Other Names: Transcranial Magnetic Stimulation,; High frequency repetitive TMS
  Arms: High frequency rTMS
Device: Placebo Stimulation — Sham Stimulation (Sham coil):right DLPFC continuous TBS, followed by left DLPFC intermitted TBS each with 50 Hz, together 1200 Stimuli, 80% motorthreshold
  Other Names: Transcranial Magnetic Stimulation; Sham Stimulation
  Arms: Placebo Stimulation

SUMMARY:
Repetitive Transcranial Magnetic Stimulation (rTMS) as well as Theta- Burst Stimulation of the frontal cortex are used to modulate the neuronal excitability in patients with depression. In the proposed study we investigate whether high frequent rTMS or Theta-Burst Stimulation of the DLPFC is more effective in patients with a depressive episode.

DETAILED DESCRIPTION:
Depression is a common mental disorder that presents with depressed mood, loss of interest, feelings of guilt or low self-worth, disturbed sleep or appetite, low energy, and poor concentration. These problems can become chronic or recurrent and lead to substantial impairments in an individual's ability to take care of his or her everyday responsibilities, at its worst, depression can lead to suicide.Depression can be reliably diagnosed in primary care. Antidepressant medications and brief, structured forms of psychotherapy are effective for 60-80 % of those affected and can be delivered in primary care.

In patients with depression the cerebral metabolism is deranged in some specific areas such as hypoexcitability in frontal cortical areas. High-frequency rTMS of the dorsolateral prefrontal cortex (DLPFC) has been investigated for the treatment of hypoexcitability disorders. Pilot data indicate that the mild effects of the rTMS could be increased by a special kind of TMS, the Theta-burst stimulation. In the proposed study we investigate whether high frequent rTMS or Theta-Burst Stimulation of the DLPFC is more effective in patients with a depressive episode.

ELIGIBILITY:
Inclusion Criteria:

* Episode of depression (unipolar or bipolar)( ICD-10)
* Female or male between 18 and 70 years
* Skills to participate in all study procedures
* 18 or more points in the Hamiliton rating scale or depression
* Stable antidepressant drugs
* Written informed consent

Exclusion Criteria:

* Clinically relevant unstable internal or neurological comorbidity
* Evidence of significant brain malformations or neoplasm, head injury
* Cerebral vascular events
* Neurodegenerative disorders affecting the brain or prior brain surgery
* Metal objects in and around body that can not be removed
* Pregnancy
* Alcohol or drug abuse
* Epilepsy or a pathological EEG
* Heart pacemaker
* High dose tranquillizers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-04; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Change in depression severity measured by the 21-item Hamilton Depression Rating Scale (Baseline versus end of treatment/ day 19) | 19 days

SECONDARY OUTCOMES:
Change in the Beck Depression Inventar, the Clinical Global Impression Scale, the Global Assessment of Functioning scale, the Alertness (Baseline versus end of treatment/ day 19, follow-up I/ day 47, follow-up II/ day 75) | 75 days
Number of responders (response = decrease of the Hamilton Depression rating scale for at least 50%) (Baseline versus end of treatment/ day 19, follow-up I/ day 47, follow-up II/ day 75) | 75 days

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Langguth, MD, Principal Investigator — University of Regensburg- Dept. of Psychiatry; Michael Landgrebe, MD, Principal Investigator — University of Regensburg, Dept. of Psychiatry; Julia Burger, MD, Principal Investigator — University of Regensburg- Dept. of Psychiatry
Locations (1):
- University of Regensburg- Dept of Psychiatry, Regensburg, Bavaria, Germany